CLINICAL TRIAL: NCT01191099
Title: Comprehensive Analysis of Hypoxia in Prostate Cancer: Diagnostic Markers and Prognostic Significance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Record Dates: First submitted 2010-08-25; First posted 2010-08-30 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prostate
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pimonidazol — 0.5gm/m2 Pimonidazol i.v. 16-24 hours before prostatectomy
  Other Names: Hypoxyprobe

SUMMARY:
A single-center cohort study to identify uni- and multivariate associations between marker gene expression and clinico-pathological parameters for the detection of robust and novel prognostic tools in prostate cancer

DETAILED DESCRIPTION:
1. To perform a large scale assessment of tissue hypoxia by pimonidazole and hypoxia marker gene expression in human prostate cancers
2. To characterize expression and hypoxia/HIF-responsiveness of myoglobin, cytoglobin, α-hemoglobin in prostate tumors and cell lines
3. To identify uni- and multivariate associations between marker gene expression and clinico-pathological parameters for the detection of robust and novel prognostic tools in prostate cancers

ELIGIBILITY:
Inclusion criteria:

* Patients with biopsy-proven adenocarcinoma of the prostate who are to be treated with radical prostatectomy at the Department of Urology, University Hospital of Zurich
* Written informed consent

Exclusion criteria:

* Metastatic prostate cancer
* Contraindications to the class of investigational product under study, e.g. known hypersensitivity or allergy to the investigational product
* Severe heart or lung disease
* Severe liver or kidney dysfunction
* Severe stridor
* Distant metastases
* Concurrent treatment for other malignant disease
* Prior hormonal therapy or radiotherapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with biopsy-proven adenocarcinoma of the prostate who are to be treated with radical prostatectomy at the Department of Urology, University Hospital of Zurich
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2020-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Michael Müntener, MD, Principal Investigator — University Hospital Zurich, Division of urology
Locations (1):
- University Hospital Zürich, Zurich, Switzerland